CLINICAL TRIAL: NCT04659564
Title: Clinical Evaluation of a Novel Wearable Compression Technology in the Treatment of Lymphedema, An Open-Label Controlled Study
Acronym: DAYSPRING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koya Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCT001
Record Dates: First submitted 2020-11-10; First posted 2020-12-09 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer Related Lymphedema; Lymphedema of Upper Arm; Lymphedema; Quality of Life
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Breast-cancer related lymphedema (BCRL) (Other)
  Interventions: Device: User of Dayspring device

INTERVENTIONS:
Device: User of Dayspring device — The Dayspring™ device is a novel FDA-cleared wearable solution that is portable and easy-to-use sequential compression system.

SUMMARY:
An open-label study to clinically assess a novel wearable advanced compression technology (Dayspring™) undertaken to determine if potential barriers to lymphedema self-care were effectively addressed. The Dayspring™ device is a novel FDA-cleared wearable solution that is portable and easy-to-use sequential compression system. The following endpoints are examined:

1. Improvement in QoL in subject with upper-extremity edema after 28 days as measured by the LYMQOL disease-specific validated assessment tool.
2. Arm volume maintenance or improvement as measured prior to and after 28 days of device use.
3. Safety as assessed by reported adverse events
4. Patient satisfaction as measured by visual analog scale (VAS) and survey at the end of the study; and
5. Adherence to therapy as measured with a smart phone app.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Willing to sign the informed consent and deemed capable of following the study protocol
* Subjects must have a diagnosis of primary or secondary unilateral or bilateral upper extremity edema

Exclusion Criteria:

* Individuals with a history or presence of a systemic disorder or condition that could place the patient at increased risk from sequential compression therapy
* Inability or unwillingness to participate in all aspects of study protocol and/or inability to provide informed consent
* Patients with exam results that would prevent safe and effective use of the study device (cellulitis, open-wounds, healing-wounds, etc.)
* Diagnosis of active or recurrent cancer, or less than 3 months at the time of initial evaluation from the completion of chemotherapy, radiation therapy or primary surgery for the treatment of cancer
* Diagnosis of Acute infection (in the last two weeks)
* Diagnosis of acute thrombophlebitis (in last 2 months)
* Diagnosis of peripheral arterial disease (PAD): PAD is defined as an Ankle Brachial Index (ABI), of 0.7 or lower
* Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 6 months
* Diagnosis of pulmonary edema
* Diagnosis of congestive heart failure (uncontrolled)
* Diagnosis of chronic kidney disease
* Diagnosis of epilepsy
* Patients with poorly controlled asthma
* Any condition where increased venous and lymphatic return is undesirable
* Women who are pregnant, planning a pregnancy or nursing at study entry
* Participation in any clinical trial of an investigational substance or device during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
LYMQOL (LYMphedema Quality of Life) | 28 days
  The Lymphedema Quality of Life Questionnaire (LYMQOL), a validated disease-specific QoL tool, was also administered at baseline and at day 28. Overall QoL is scored on a single item by the patient on a scale of 1-10.
Arm Volume Maintenance or Improvement | 28 days
  Limb volume measurement was performed by using a calibrated tape measure to measure circumference from the wrist and the ulnar styloid process and at 4cm increments to the axilla. Measurements were taken for both upper extremities. If both extremities exhibited edema, a study arm was designated for treatment. Measurements were taken by the same investigator throughout the study. Volume was calculated based on cylindrical segment analysis.
Safety/AEs | 28 days
  As assessed by reported adverse events
Therapy adherence tracking | 28 days
  Therapy adherence tracked via the mobile app linked to the Dayspring™ device.

SECONDARY OUTCOMES:
Patient survey | 28 days
  A visual analog scale (VAS) and study survey were administered at the end of the study to measure patient satisfaction (day 28). The six-item questionnaire was used to document the time of day the device was used, if daily activities were supported during use, function, and symptoms. All were measured on a scale from 1-5. The VAS was administered to previous users of pneumatic compression devices to assess preference and likelihood to recommend to others with lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, MD, Principal Investigator — Medical Advisor
Locations (2):
- United States (2):
  - PT works, Los Altos, California
  - Ginger-K Lymphedema & Cancer Center, Morgan Hill, California